CLINICAL TRIAL: NCT01230684
Title: Comparison of Contrast Enhanced Ultrasound and the Gold Standard Computed Tomographic Angiography in Detection of Endoleak Following Endovascular Abdominal Aortic Aneurysm Repair.
Brief Title: Contrast Enhanced Ultrasound vs. Computed Tomographic Angiography in the Detection of Endoleaks Following AAA Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan Eliason, MD, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00038554; Internal Grant Award (Other Grant/Funding Number: G009310/Cardiovascular Center)
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Endograft Implantation to Repair Abdominal Aortic Aneurysm
Keywords: CEUS; Endoleaks; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Endoleak; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoleak imaging (Other): In the single arm all participants are recieving both imaging techniques; CEUS and CTA
  Interventions: Procedure: Contrast Enhanced Ultrasound (Contrast Agent: OptisonTM)

INTERVENTIONS:
Procedure: Contrast Enhanced Ultrasound (Contrast Agent: OptisonTM) — The contrast agent will be prepared using a single, 3 mL vial of Optison and 57 mL saline combined in a sterile syringe. Contrast will be set to deliver a continuous infusion at 4 mL/min, via peripheral access. In the event that the above description of the administration of Optison is not adequate for lumen flow contrast enhancement the PI or Co-I will direct the study team to proceed to the secondary administration procedure. This will be done by the following: 0.5 mL of Optison will be injected into a peripheral vein. This may be repeated for further contrast enhancement as needed. The maximum total doses should not exceed 5.0 mL in any 10 minute period nor exceed 8.7 mL in any one patient study. We will follow the insert package dose. We will not not exceed 5.0 or 10 minutes or 8.7ml per patient (this will include the 0.5mL for initial). Therefore, no more that 8.2mL will given in this second administration procedure.

SUMMARY:
The purpose of the study is to compare two different types of imaging techniques to identify endoleaks. Following the endovascular procedure, subjects are seen at one month to have computed tomographic angiography (CTA) to confirm the graft is not leaking (endoleak). CTA is the standard imaging technique used to identify endoleaks. This study will investigate if the image technique color duplex ultrasound with contrast enhanced ultrasound (CEUS) is a good tool to identify endoleaks too.

DETAILED DESCRIPTION:
Background:

Abdominal aortic aneurysms (AAAs) continue to be a leading cause of death in older age groups. In the 60-85 year-old population, AAA represents the 14th-leading cause of death. Federal funding through Medicare has been allocated for early detection using abdominal ultrasound screening programs. Despite these more aggressive screening programs and concerted efforts by surgeons for timely repair, the incidence of ruptured AAA has continued to increase.

Endovascular aneurysm repair (EVAR) has been the most common type of repair since 2006. Multiple studies reflecting decreased perioperative morbidity and mortality over open repair make this an attractive option for patients. EVAR requires more intensive follow-up than standard open surgical repair, however. Secondary interventions are more common to maintain "seal" of the endograft within the aorta and subsequent exclusion of the aneurysmal component.

The term endoleak is specific to EVAR, and describes the primary means by which endografts fail. Type I endoleaks occur because of inadequate graft seal proximally or distally, resulting in perigraft flow and aneurysm sac pressurization. Type II endoleaks occur when branch arteries arising from the aneurysmal aorta back-bleed into the aneurysm sac due to collateral flow. Type III endoleaks occur when flow persists between segments of a modular graft. Type IV endoleaks occur when flow persists through endograft material (graft porosity). Type V endoleaks have also been called "endotension", and occur when pressurization of the sac occurs in the absence of any demonstrable endoleak. Type I and Type III endoleaks are most concerning for rupture, although persistent Type II endoleaks can also lead to aneurysm rupture and premature death.

The most common method of EVAR follow-up is computed tomographic angiography (CTA). These studies allow accurate measurement of aneurysm sac diameters and volumes. They also are highly sensitive and specific for endoleaks. Type II endoleaks are treated if they remain persistent and are present in the setting of aneurysm sac enlargement. Type I and III endoleaks are immediately treated when identified. Type IV endoleaks are rarely seen with current endograft technology.

Study Objectives:

The purpose of the current study is to compare routine postoperative surveillance by CTA with color duplex ultrasound and contrast enhanced ultrasound (CEUS) for the detection of endoleaks.

Study Design

This is a pilot study comparing the imaging techniques of CTA to CEUS in 25 patients undergoing EVAR at their one month post endograft surveillance. The one month standard follow-up will be used for comparing techniques as this will yield the highest number of endoleak positive patients. Patients will complete a color duplex examination in conjunction with CEUS using the FDA approved ultrasound contrast agent OptisonTM (Perflutren Protein Type A Microspheres for Injection, USP). Following ultrasonographic evaluation, study patients will undergo routine CTA.

Eligible subjects will be asked to participate in the trial following post-op day number 1 from their endovascular procedure. Study participation is ~30 days (+ 7 days).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and greater
* Men or postmenopausal/non-pregnant women
* Abdominal aortic aneurysm successfully repaired by endograft deployment
* Creatinine < 2.0 mL
* Planned CTA follow-up

Exclusion Criteria:

* Subjects with known or suspected hypersensitivity to blood, blood products, or albumin.
* Subjects unable/unwilling to give informed consent
* Unable to complete post-operative imaging studies
* Subjects identified to have a cardiac shunt by TTE
* Subjects with hepatic or respiratory disease
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Patient diagnosed with endoleak via CEUS and confirmed by CTA | 30 days postoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: Jon Eliason, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States